CLINICAL TRIAL: NCT00972998
Title: An Open Label Study to Examine the Effect of Coated Phenylephrine Suppositories on Anal Pressure in Healthy Subjects
Brief Title: Study to Examine the Effect of Coated Phenylephrine Suppositories on Anal Pressure in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Michael Shapiro MD, Gastroenterology Dept, Asaf Harofe Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RDD 105
Record Dates: First submitted 2009-08-17; First posted 2009-09-09 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Incontinence
Keywords: anal sphincter pressure; phenyephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy individuals (Experimental)
  Interventions: Drug: Phenyephrine

INTERVENTIONS:
Drug: Phenyephrine — Phenyephrine coated suppositories

SUMMARY:
This is an open label, dose-finding study. Approximately 8 healthy subjects will be participating in this study.

A screening will be used to determine subject suitability for inclusion in the trial. Subjects who meet all inclusion criteria and none of the exclusion criteria will enter a one day treatment period. During this period, 4 anal manometric studies will take place. Study medication (Coated Phenylephrine suppositories at various doses) will be administered at pre-determined intervals.

DETAILED DESCRIPTION:
This is an open label, dose-finding study. Approximately 8 healthy subjects will be participating in this study. A screening will be used to determine subject suitability for inclusion in the trial. Within one week after the screening visit, subjects who meet all inclusion criteria and none of the exclusion criteria will enter a one day treatment period. During this period, 4 anal manometric studies will take place. Study medication (Coated Phenylephrine suppositories at various doses) will be administered at pre-determined intervals. During the study, blood samples will be obtained for plasma Phenylephrine analysis.After determining baseline resting anal pressure with a manometric test, coated Suppositories will be administered intra rectally. Subjects will take rectally a total of 1 Coated Suppository per study. 60, 120 and 240 minutes after the coated suppository insertion amnometric studies will be performed: The first 2 subjects in the study will receive 40 mg phenyephrine coated suppositories. If significant (> 15%) increase in the resting anal pressure will occur with this dose, the rest of the study subjects will receive the same dose. If the raise in the resting anal pressure will not be significant AND no adverse events was observed, than the following subjects will receive 80 mg phenylehprine coated suppositories.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female subjects 18 to 55 years of age.

Exclusion Criteria:

* Active or chronic disease.
* In need of chronic use of medication, with the exception of birth control medications.
* Currently uses medication for acute illness.
* Has used, in the last four weeks, drugs that may affect blood coagulation, such as Aspirin, Warfarin, Sintrom, Enoxaparin, Nadroparin, Heparin, Clopidogrel, Ticlopidine.
* Has upon physical examination a rectal deformation or signs of rectal disease such as fissure, bleeding hemorrhoids, fistula., infection or space occupying lesion.
* Receipt of any investigational treatment (drug or device) within 90 days prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter is change in Resting Anal Pressure from baseline. | 8 hours

SECONDARY OUTCOMES:
The ratio of change in anal pressure to plasma Phenylephrine level. | 8 hours
The ratio of change in anal pressure to change in blood pressure. | 8 hours
The ratio of change in anal pressure to change in heart rate. | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Shapiro, MD, Principal Investigator — Dept of gastroeneterology, asaf harofe medical center
Locations (1):
- Dept of Gastroeneterology, Asaf Harofe Medical Center, Zrifin, Israel